CLINICAL TRIAL: NCT03944746
Title: Assessment of an Orthopedic Surgery Rotation on Musculoskeletal Competency in Emergency Medicine Residency Training
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jared L. Cohen (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jared L. Cohen, Emergency Medicine Physician, San Antonio Military Medical Center
Organization: San Antonio Military Medical Center (U.S. Federal Agency)
Other Study IDs: MCHE-CI; 32 CFR 219.102(d)
Record Dates: First submitted 2019-05-03; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Educational Problems; Orthopedic Disorder; Emergencies
Keywords: Emergency Department Education
MeSH Terms: conditions — Musculoskeletal Diseases; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SAMMC Emergency Medicine Residents: Emergency Medicine Residents from San Antonio Military Medical Center in San Antonio, Texas.
  Interventions: Other: Education Curriculum
- University Hospital Emergency Medicine Residents: Emergency Medicine Residents from University Hospital in San Antonio, Texas.
  Interventions: Other: Education Curriculum

INTERVENTIONS:
Other: Education Curriculum — Different educational curriculums were applied to each cohort

SUMMARY:
Patient commonly present with orthopedic injuries in the emergency department. Musculoskeletal education has not historically been emphasized in American medical schools, and the effectiveness of an orthopedic surgery rotation has not been well studied in emergency medicine (EM) training. Competency in musculoskeletal education has been tested previously with a validated instrument, the basic competency exam (BCE), to assess baseline knowledge in primary care and emergency physicians.

Residents from 2 different EM residency training programs will be given the BCE to determine baseline musculoskeletal knowledge prior to their orthopedic surgery rotations. A post-test BCE will be given to the residents from both EM training programs upon completion of their orthopedic surgery rotation and compared.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medicine Residents at either San Antonio Military Medical Center or University Hospital

Exclusion Criteria:

* Not emergency medicine residents at the inclusion sites.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population is whoever is an emergency medicine resident at the programs listed previously.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-11-13 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in performance on the orthopedic basic competency exam | Assessed initially by taking the exam before completing a one month orthopedic rotation. The same exam is taken at the completion of the orthopedic rotation. The two test results are compared to each other between each individual and residency program.
  The orthopedic basic competency exam is a validated scoring system meant to assess the learner's ability to evaluate both emergent and common orthopedic pathology. It is a 25 question test, and the test-taker will receive a score between 0 and 25.

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio Military Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No